CLINICAL TRIAL: NCT01261390
Title: A Planning Study: Sleep Apnea Intervention for Cardiovascular Disease Reduction
Brief Title: Sleep Apnea Intervention for Cardiovascular Disease Reduction
Acronym: BestAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Susan Redline, Professor and Senior Physician of Sleep Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P002671
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea; Heart Disease; Risk factors for heart disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Conservative Medical Therapy (CMT) (Placebo Comparator): All participants will meet with a research assistant who will provide ~30 minutes of instruction on sleep hygiene and healthy lifestyle guidelines. Each subject's sleep routine will be reviewed with the aim to identify appropriate bed and wake times that provide a consistent schedule and allow for at least 7 hours of time in bed per night. Habits that may impact sleep, such as alcohol consumption, tobacco use, and exercise close to bedtime will be reviewed with appropriate guidance on how to minimize sleep disrupting exposures. Subjects will be provided external nasal dilator strips (Breath Right®) and advised on how to maximize sleep time in a non-supine position using bed elevation, wedge pillows and/or objects affixed to the back of their night clothes as appropriate.
  Interventions: Behavioral: Conservative Medical Therapy (CMT)
- Sham PAP (Sham) (Sham Comparator): In addition to receiving CMT, participants in this treatment arm will receive a sham-CPAP unit. Sham devices look like active PAP devices, however, the exhalation port is increased and an orifice-resistor is inserted between the pump and tubing, creating a marginal pressure. A heated humidifier will be provided with this device and PAP masks will be fit and provided following the same procedures as for the active PAP arms.
  The treatment visit schedule is outlined below.
  1. PAP Initial Set-Up
  2. 1-week follow up
  3. 1-month follow up
  4. 3-month follow up
  5. 6-month follow up
  6. 9-month follow up (will not occur if on a 6-month follow-up protocol)
  It is estimated that each in-person follow-up adherence visit with the PAP specialist would last ~30 minutes.
  Interventions: Behavioral: Conservative Medical Therapy (CMT); Device: Sham PAP (Sham)
- Active PAP with RT Support (Active-Beh) (Active Comparator): In addition to receiving CMT, participants will receive active-PAP. The treatment visit schedule is outlined below.
  1. PAP Initial Set-Up
  2. 1-week follow up (FU)
  3. 1-month FU
  4. 3-month FU
  5. 6-month FU
  6. 9-month FU (12-month follow-up protocol only)
  All visits will take place with a PAP specialist. All follow-up visits will be anchored to the initial PAP set-up visit. At these visits, using the available data from the PAP monitor, the PAP specialist will discuss PAP use, mask leaks, and residual AHI to assist with troubleshooting. Adjustments to equipment would be performed as needed to improve adherence. Each follow-up visit with the PAP specialist will last 30 minutes.
  Interventions: Behavioral: Conservative Medical Therapy (CMT); Device: Active PAP with RT Support (Active-Beh)
- Active PAP with Behavioral Modification (Active+Beh) (Active Comparator): In addition to receiving CMT and active-PAP, participants will have behavioral intervention sessions to promote PAP adherence. The treatment visit schedule is outlined below:
  Visits with Behavioral Interventionist (in addition to active-PAP treatment visits):
  1. PAP Initial Set-Up (in-person, 1-hr)
  2. 1-week follow-up (FU) (in-person, 1-hr)
  3. 1-month FU
  4. 2-month FU
  5. 3-month FU
  6. 5-month FU
  7. 8-month FU (12-month follow-up protocol only)
  All follow-up visits will be anchored to the initial PAP set-up visit. PAP treatment visits will occur as outlined in the active-PAP arm.
  All behavioral intervention visits will be 30-min phone calls, unless otherwise noted. The intervention will be based on social cognitive theory and feedback concerning adherence with targeted problem solving training.
  Interventions: Behavioral: Conservative Medical Therapy (CMT); Device: Active PAP with Behavioral Modification (Active+Beh)

INTERVENTIONS:
Behavioral: Conservative Medical Therapy (CMT) — All participants will meet with a research assistant who will provide 30 minutes of instruction on sleep hygiene and healthy lifestyle guidelines. Each subject's sleep routine will be reviewed with the aim to identify appropriate bed and wake times that provide a consistent schedule and allow for at least 7 hours of time in bed per night. Habits that may impact sleep, such as alcohol consumption, tobacco use, and exercise close to bedtime will be reviewed with appropriate guidance on how to minimize sleep disrupting exposures. Subjects will be provided external nasal dilator strips (Breathe Right®) and advised on how to maximize sleep time in a non-supine position using bed elevation, wedge pillows and/or objects affixed to the back of their night clothes as appropriate.
  Other Names: Breathe Right® external dilator strips
Device: Sham PAP (Sham) — In addition to receiving CMT, participants in this treatment arm will receive a sham PAP unit. Sham devices look like active PAP devices, however, the exhalation port is increased and an orifice-resistor is inserted between the pump and tubing, creating a marginal pressure. A heated humidifier will be provided with this device and PAP masks will be fit and provided following the same procedures as for the active-PAP arms.
  Other Names: REMstar Pro M Series (Philips-Respironics); S9 (ResMed)
  Arms: Sham PAP (Sham)
Device: Active PAP with RT Support (Active-Beh) — In addition to receiving CMT, participants will receive active-PAP and meet with a PAP-specialist . The CPAP specialist would meet with the participant in person throughout the course of the study (set-up, 1-week, 1-month, 3-month, 6-month, and 9-month). Using the available data from the PAP monitor, the PAP specialist will discuss PAP use, mask leaks, and residual AHI to assist with troubleshooting. Adjustments to equipment would be performed as needed to improve adherence. It is estimated that each in-person follow-up adherence visit with the PAP-specialist would last 30 minutes.
  Other Names: REMstar Pro M Series (Philips-Respironics); S9 (ResMed)
  Arms: Active PAP with RT Support (Active-Beh)
Device: Active PAP with Behavioral Modification (Active+Beh) — In addition to receiving CMT and active-PAP, participants will meet with a behavioral interventionist in addition to PAP-specialist visits. Participants also would speak with the behavioral interventionist over the course of the study (set up, 1-week, 3-week, 1-month, 2-months, 3-months, 5-months and 8-months). The duration of the first 2 behavioral intervention sessions are estimated to be 1-hour long, with subsequent 30-minutes intervention sessions. The intervention will be based on social cognitive theory and feedback concerning adherence with targeted problem solving training.
  Other Names: REMstar Pro M Series (Philips-Respironics); S9 (ResMed)
  Arms: Active PAP with Behavioral Modification (Active+Beh)

SUMMARY:
Moderate to severe sleep apnea (a high number of breathing pauses on a sleep study) is a common health problem that is often associated with loud snoring and sleepiness.The medical term for this problem is obstructive sleep apnea (OSA). People with OSA often have an increased risk for developing heart disease or may already have a diagnosis of heart disease.

A clinical research study is being conducted at Brigham and Women's Hospital (BWH) and Beth Israel Deaconess Medical Center (BIDMC) to compare the effects of continuous positive airway pressure (CPAP) to conservative medical therapy with participation in one of four groups:

1. Active-PAP Therapy Group (Active-Beh or Active+Beh): Will receive standard medical treatment for sleep apnea with active-PAP. Participants will be randomized to either:

   1. Active-Pap with respiratory therapist visits only
   2. Active-Pap with respiratory therapist visits and cognitive behavioral therapist visits.
2. Alternative PAP Group (Sham): Will receive lower air delivery level than active-PAP therapy group. Will also have meetings with respiratory therapist.
3. Conservative Medical Therapy Group (CMT)*: Will receive a free supply of nasal strips for the duration of their treatment period (either 6 months or 12 months) and follow healthy sleep hygiene guidelines for how to change sleep habits to minimize incidences of apneas (breathing disturbances during sleep). Frequent follow-up support with research coordinator.

A sleep doctor or cardiologist will have indicated that a potential participant is an appropriate candidate to receive PAP or CMT as acceptable approaches to treat his/her sleep apnea. Participants will be recruited between the ages of 45-75 years who have diagnosed heart disease or between 55-75 years for those who have risk factors for developing heart disease.

This is a 6-12 month study** to evaluate alternative ways to address the potential for OSA treatment to reduce heart disease and to identify those features that would strengthen a later, large-scale randomized controlled trial.

We will test the hypothesis that active treatment for OSA with CPAP reduces CVD morbidity and mortality.

*All randomized participants will be given conservative medical therapy (CMT).

**For those randomized after December 31, 2012, follow-up assessment will only be 6 months long

DETAILED DESCRIPTION:
In this pilot randomized controlled trial, we will assess the effectiveness of CPAP therapy to reduce the burden of cardiovascular disease (CVD) and CVD risk factors in patients with moderate to severe obstructive sleep apnea (OSA) presenting to a sleep disorders clinic. A total of 700 patients with a new diagnosis of moderate to severe OSA will be recruited from BWH-affiliated sleep disorder clinics, BWH, Massachusetts General Hospital (MGH), and Faulkner Hospital Cardiology Clinics (and similar specialized clinics seeing patients with cardiovascular risk factors, such as endocrinology and hypertensive clinics), Beth Israel Deaconess Medical Center and Joslin Diabetes Center. After completing a 2 week run-in period, randomized participants (approximately 150 participants will be randomized) will undergo baseline and 6 month assessments of key study exposure and outcome variables.

Participants will be randomized after completion of Baseline visit. The treatment arms are as follows:

The active arms are:

1. Active-PAP treatment delivered using standard respiratory therapist (RT) adherence education and support. (Active-Beh)
2. Active-PAP treatment administered using adherence education and support delivered by a RT and enhanced by a behavioral promotion intervention. (Active+Beh)

The control arms are:

1. Conservative Medical Therapy (CMT)
2. Sham-PAP (Sham)

Participants randomized before December 31, 2012 (n=108) also will undergo 12 month follow-up assessments. Participants will be offered a 12 month supervised conservative medical therapy (CMT) program for OSA over the duration of the study intervention. Subjects would be contacted at bimonthly intervals by alternating phone and office visits to assess safety, identify adverse events, identify health care utilization, and reinforce protocol adherence. At 6 and 12 months, study outcomes will be reassessed by collecting data from sources.

Patients randomized after December 31, 2012 (n=61) will undergo only 6 months of follow-up assessment. Participants will be offered a 6 month supervised conservative medical therapy (CMT) program for OSA over the duration of the study intervention. Subjects would be contacted at bimonthly intervals by alternating phone and office visits to assess safety, identify adverse events, identify health care utilization, and reinforce protocol adherence. At 6 months, study outcomes will be reassessed by collecting data from sources.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive apnea hypopnea index (AHI) ≥ 15
* Age 45-75 years, or 55 to 75 yrs if without established Cardiovascular Disease (CVD)
* Ability to provide informed consent, with the patient and physician acknowledging accepting uncertainty on the role of PAP in CVD prevention.
* Established CVD,or having diabetes mellitus, defined by one or more of the following:

  1. Prior myocardial infarction
  2. Coronary artery revascularization procedure (≥4 months before study entry)
  3. Angiographically documented stenosis (>70%) of a major coronary artery
  4. Prior ischemic stroke without major functional impairment
  5. Diabetes mellitus treated with medication or ≥ 2 fasting glucose levels ≥ 126 mg/dl

OR

Three or more of the following established CVD risk factors:

1. Hypertension treated with medications or systolic BP > 140 or diastolic BP > 90 on ≥ 2 occasions
2. Male sex
3. BMI ≥ 30
4. Total cholesterol > 240 mg/dl or LDL cholesterol > 160 mg/dl or HDL < 45 mg/dl
5. > 10 pack years of smoking

Exclusion Criteria:

* Diagnosed heart failure with known cardiac ejection fraction of < 35% or New York Heart Association (NYHA) class 3 or 4 status
* Less than 4 months since myocardial infarction (MI), stroke or revascularization procedure
* Poorly controlled hypertension (>170/>100)
* Prior stroke with functional impairment interfering with ability to complete the protocol
* Severe uncontrolled medical problems or medications that may influence measurements or impair ability to participate in the study exams (e.g. oral steroids; chronic opioid use; self- reported chronic kidney disease or, if measured, creatinine > 2.5 mg/dl or glomerular filtration rate (GFR) < 30; anemia with Hgb < 10, etc.)
* Resting oxygen saturation < 90% or nocturnal oxygen saturation <85% for > 10% of the sleep period;
* Use of prescribed PAP for sleep apnea within the prior 2 years
* Report of inability to spend >6 hrs in bed
* Any use of prescribed PAP for sleep apnea
* Severe sleepiness defined by an Epworth Sleepiness Score of >14 or report of falling asleep driving in the prior 2 years
* Working as a professional driver
* Low risk related to having sleep apnea defined by a Berlin Score < 2
* Central sleep apnea, with >50% of respiratory events classified as central apneas
* Refusal to consider PAP use after an initial split-night PAP study (pre-randomization)
* Concurrent involvement in another research study that will result in a conflict as determined by study doctors

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2011-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Murray Mittleman, MD, DrPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zhao YY, Wang R, Gleason KJ, Lewis EF, Quan SF, Toth CM, Song Y, Morrical M, Rueschman M, Mittleman MA, Redline S. Effect of continuous positive airway pressure treatment on ambulatory blood pressures in high-risk sleep apnea patients: a randomized controlled trial. J Clin Sleep Med. 2022 Aug 1;18(8):1899-1907. doi: 10.5664/jcsm.10012. PMID 35459446
- [Derived] Reid ML, Gleason KJ, Bakker JP, Wang R, Mittleman MA, Redline S. The role of sham continuous positive airway pressure as a placebo in controlled trials: Best Apnea Interventions for Research Trial. Sleep. 2019 Aug 1;42(8):zsz099. doi: 10.1093/sleep/zsz099. PMID 31116848
- [Derived] Bakker JP, Wang R, Weng J, Aloia MS, Toth C, Morrical MG, Gleason KJ, Rueschman M, Dorsey C, Patel SR, Ware JH, Mittleman MA, Redline S. Motivational Enhancement for Increasing Adherence to CPAP: A Randomized Controlled Trial. Chest. 2016 Aug;150(2):337-45. doi: 10.1016/j.chest.2016.03.019. Epub 2016 Mar 24. PMID 27018174
- [Derived] Yaggi HK, Mittleman MA, Bravata DM, Concato J, Ware J, Stoney CM, Redline S. Reducing cardiovascular risk through treatment of obstructive sleep apnea: 2 methodological approaches. Am Heart J. 2016 Feb;172:135-43. doi: 10.1016/j.ahj.2015.07.033. Epub 2015 Sep 11. PMID 26856225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial recruitment was limited to patients with sleep apnea identified through clinical sleep programs of Brigham and Women's Hospital (BWH) and Beth Israel Deaconess Medical Center (BIDMC). Recruitment later expanded to include patients presenting to cardiology and diabetes clinics. Recruitment began on April 2011 and ended on June 2013.
Pre-assignment Details: Patients with no sleep study were provided a portable sleep monitor to measure the severity (if any) of obstructive sleep apnea (OSA). If tests shows moderate to severe OSA, patients were asked to wear a positive airway pressure (PAP) mask with no pressure for 2 weeks. Those with proven adherence during this time were scheduled for a baseline visit
Groups:
- Active PAP With RT Support (Active-Beh): In addition to receiving CMT, participants will receive active-PAP and meet with a PAP-specialist . The PAP specialist would meet with the participant in person throughout the course of the study (set-up, 1-week, 1-month, 3-month, 6-month, and 9-month). Using the available data from the PAP monitor, the PAP specialist will discuss PAP use, mask leaks, and residual apnea hypopnea index (AHI) to assist with troubleshooting. Adjustments to equipment would be performed as needed to improve adherence. It is estimated that each in-person follow-up adherence visit with the PAP-specialist would last 30 minutes.
Period: Overall Study
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Started | 44 (15 of the 44 participants only had to complete a 6-month follow-up assessment.) | 42 (15 of the 42 participants only had to complete a 6-month follow-up assessment.) | 42 (16 of the 42 participants only had to complete a 6-month follow-up assessment.) | 41 (15 of the 41 participants only had to complete a 6-month follow-up assessment.)
6-Month Visit | 37 (For 14 of the 30 participants in this arm, this was their final visit.) | 34 (For 12 of the 34 participants in this arm, this was their final visit.) | 34 (For 16 of the 34 participants in this arm, this was their final visit.) | 32 (For 14 of the 32 participants in this arm, this was their final visit.)
12-Month Visit | 23 | 21 | 19 | 19
Completed | 37 (14 of the 37 participants that completed the study in this arm were under the 6-Month protocol.) | 33 (12 of the 33 participants that completed the study in this arm were under the 6-Month protocol.) | 35 (16 of the 35 participants that completed the study in this arm were under the 6-Month protocol.) | 33 (14 of the 33 participants that completed the study in this arm were under the 6-Month protocol.)
Not Completed | 7 | 9 | 7 | 8
Not completed — Significant Concurrent Illness | 1 | 0 | 1 | 0
Not completed — Dissatisfaction with Treatment | 2 | 1 | 1 | 2
Not completed — Relocation | 0 | 1 | 0 | 0
Not completed — Loss of Interest in the Study | 3 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 6 | 5 | 6

BASELINE CHARACTERISTICS:
Population: If were not able to collect data from a participant (24-hour blood pressure monitor, echocardiogram, questionnaires, etc), we did not included them in the Baseline Analysis for that measure. This will result in different n-values for each arm.
Groups:
- Active PAP With RT Support (Active-Beh): In addition to receiving CMT, participants will receive active-PAP and meet with a PAP-specialist . The PAP specialist would meet with the participant in person throughout the course of the study (set-up, 1-week, 1-month, 3-month, 6-month, and 9-month). Using the available data from the PAP monitor, the PAP specialist will discuss PAP use, mask leaks, and residual AHI to assist with troubleshooting. Adjustments to equipment would be performed as needed to improve adherence. It is estimated that each in-person follow-up adherence visit with the PAP-specialist would last 30 minutes.
- Total: Total of all reporting groups
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh) | Total
Number analyzed (Participants) | 44 | 42 | 42 | 41 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (6.3) | 63.0 (7.5) | 63.7 (7.3) | 63.6 (8.2) | 63.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 14 | 14 | 59
  Male | 32 | 23 | 28 | 27 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3 | 6
  Not Hispanic or Latino | 43 | 41 | 41 | 38 | 163
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 3 | 2 | 11
  White | 41 | 36 | 37 | 37 | 151
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2 | 4
Cardiovascular Disease (CVD) Status [Number; unit: participants]
  CVD Risk Factors | 20 | 17 | 17 | 18 | 72
  Established CVD | 24 | 25 | 25 | 23 | 97
Diagnostic Type [Number; unit: participants]
  Full-Night | 41 | 39 | 39 | 38 | 157
  Split-Night | 3 | 3 | 3 | 3 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.4 (7.2) | 32.1 (5.7) | 30.6 (4.5) | 31.6 (5.9) | 31.7 (5.9)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 110.2 (16.1) | 112.6 (14.5) | 108.3 (12.2) | 110.6 (13.3) | 110.4 (14.1)
AHI [Mean (Standard Deviation); unit: respiratory events per hour] — AHI is an index of sleep apnea severity that combines apneas and hypopneas. The AHI is expressed as the number of respiratory events per hour.
  respiratory events per hour | 33.9 (21.8) | 31.5 (20.0) | 27.6 (12.5) | 26.8 (12.4) | 30.0 (17.4)
Baseline Resting Blood Pressure Data by Arm [Mean (Standard Deviation); unit: mmHg]
  Average Resting Systolic | 125.1 (15.3) | 123.6 (18.1) | 124.8 (19.5) | 127.5 (16.2) | 125.2 (17.2)
  Average Resting Diastolic | 70.1 (8.6) | 68.6 (8.5) | 71.2 (10.6) | 71.3 (8.9) | 70.3 (9.2)
Baseline 24-Hour Blood Pressure Data by Arm [Mean (Standard Deviation); unit: mmHg] — Blood pressure data was collected using a 24-hour ambulatory blood pressure monitor. Population: We were not able to collect 24-hour blood pressure data from all participants that completed a baseline visit.
  mmHg
    24-hour Systolic Blood Pressure: number analyzed (Participants) | 40 | 40 | 41 | 40 | 161
    24-hour Systolic Blood Pressure | 125.4 (14.3) | 128.1 (14.4) | 121.3 (10.4) | 121.8 (11.0) | 124.1 (12.8)
    Sleep Mean Arterial Pressure | 83.3 (12.4) | 84.7 (11.2) | 81.1 (8.0) | 81.5 (10.2) | 82.7 (10.6)
    24-hour Mean Arterial Pressure | 90.7 (9.8) | 92.0 (8.7) | 89.3 (6.5) | 89.2 (7.4) | 90.3 (8.2)
Baseline Laboratory Measures by Arm - Triglyceride and HDL [Mean (Standard Deviation); unit: mg/dL]
  Triglyceride | 130.3 (85.8) | 125.8 (61.6) | 108.3 (57.1) | 143.8 (81.8) | 127.0 (73.2)
  HDL | 49.1 (14.9) | 50.0 (12.2) | 55.7 (16.9) | 47.4 (12.9) | 50.5 (14.6)
Baseline Laboratory Measures by Arm - CRP [Mean (Standard Deviation); unit: mg/L] — Population: We were not able to collect C-Reactive Protein (CRP) values from all participants that completed a baseline visit.
  mg/L
    number analyzed (Participants) | 44 | 42 | 42 | 40 | 168
    (all) | 3.9 (9.0) | 5.6 (17.6) | 4.5 (10.4) | 3.0 (2.7) | 4.3 (11.2)
Baseline Echocardiogram Measures by Arm - Pulse Wave Velocity [Mean (Standard Deviation); unit: m/s] — Population: We were not able to collect pulse wave velocity values from all participants that completed a baseline visit.
  m/s
    number analyzed (Participants) | 34 | 34 | 39 | 38 | 145
    (all) | 9.6 (2.1) | 9.7 (2.4) | 8.6 (1.8) | 9.4 (1.8) | 9.3 (2.1)
Baseline Echocardiogram Measures by Arm - Augmentation Index [Mean (Standard Deviation); unit: percent of central pulse pressure] — Population: We were not able to collect augmentation index values from all participants that completed a baseline visit.
  percent of central pulse pressure
    number analyzed (Participants) | 41 | 38 | 41 | 39 | 159
    (all) | 30.6 (9.6) | 30.2 (9.7) | 29.8 (9.3) | 29.8 (8.7) | 30.1 (9.3)
Baseline Echocardiogram Measures by Arm - Ejection Fraction [Mean (Standard Deviation); unit: percent ejection fraction] — Population: We were not able to collect ejection fraction values from all participants that completed a baseline visit.
  percent ejection fraction
    number analyzed (Participants) | 38 | 37 | 38 | 37 | 150
    (all) | 60.2 (4.1) | 60.9 (2.7) | 60.8 (6.6) | 59.9 (4.6) | 60.5 (4.7)
Baseline Quality of Life Measures by Arm - Short Form Health Survey (SF-36) [Mean (Standard Deviation); unit: units on a scale] — The SF-36 is a patient-reported survey of patient health. The SF-36 scores range from 0-100, with lower scores indicating the more disability. Population: We were not able to collect all values from all participants that completed a baseline visit.
  units on a scale
    SF-36 Vitality Subscale: number analyzed (Participants) | 43 | 40 | 40 | 40 | 163
    SF-36 Vitality Subscale | 49.6 (10.1) | 48.0 (9.7) | 49.0 (10.4) | 48.7 (9.6) | 48.9 (9.9)
    SF-36 Emotional Subscale: number analyzed (Participants) | 43 | 40 | 40 | 40 | 163
    SF-36 Emotional Subscale | 47.9 (10.7) | 44.9 (12.3) | 48.4 (11.1) | 45.5 (12.3) | 46.7 (11.6)
    SF-36 Physical Subscale: number analyzed (Participants) | 43 | 40 | 40 | 41 | 164
    SF-36 Physical Subscale | 44.1 (10.9) | 44.3 (10.7) | 47.1 (10.0) | 44.4 (10.9) | 45.0 (10.6)
Baseline Quality of Life Measures by Arm - ESS [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness. The ESS score ranges from 0 - 24, with higher scores indicating increasing possibility of specific sleep disorders.
  We were not able to collect all values from all participants that completed a baseline visit. The following n-values apply to the respective categories below.
  CMT, n=43; Sham, n=40; Active-Beh, n=40; Active+Beh, n=41; Total, n=164
  units on a scale | 9.0 (4.9) | 8.0 (4.2) | 7.8 (4.2) | 8.4 (4.8) | 8.3 (4.5)
Baseline Quality of Life Measures by Arm - PHQ-8 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-8) is a scale intended to measure depression. The PHQ-8 score ranges from 0 - 24, with higher scores indicating increasing severity of depression. Population: We were not able to collect all values from all participants that completed a baseline visit.
  units on a scale
    number analyzed (Participants) | 42 | 40 | 38 | 40 | 160
    (all) | 5.0 (4.6) | 5.1 (4.1) | 4.7 (5.1) | 6.4 (5.6) | 5.3 (4.9)
Baseline Quality of Life Measures by Arm - SAQLI [Mean (Standard Deviation); unit: units on a scale] — The Calgary Sleep Apnea Quality of Life Index (SAQLI) is a scale intended to measure disease-specific quality of life. The SAQLI score ranges from 1 - 7, with higher scores indicating a higher quality of life. Population: We were not able to collect all values from all participants that completed a baseline visit.
  units on a scale
    number analyzed (Participants) | 43 | 41 | 41 | 41 | 166
    (all) | 4.8 (0.8) | 4.8 (0.8) | 4.9 (0.9) | 4.7 (1.0) | 4.8 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Blood Pressure at Months 6 and 12 by Pooled Arms
Description: Blood pressure data was collected using a 24-hour ambulatory blood pressure monitor. The 2 Active arms and 2 Control arms were pooled to create a 2-arm analysis. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months. Control arms and Active arms were pooled, respectively, for analysis.
Time Frame: Mean of 6- and 12-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) who had valid measurements of ambulatory blood pressure for baseline and at least one follow-up timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Control Arms (Pooled): Participants randomly assigned to either the Conservative Medical Treatment (CMT) or Sham-PAP arms.
- Active Treatment Arms (Pooled): Participants randomly assigned to either the Active-PAP + Respiratory Therapist (RT) Support or the Active-PAP + Behavioral Modification Therapy arm.
Arm/Group | Control Arms (Pooled) | Active Treatment Arms (Pooled)
Number analyzed (Participants) | 69 | 69
mmHg
  24-hour Systolic Blood Pressure: number analyzed (Participants) | 68 | 66
  24-hour Systolic Blood Pressure | 1.82 (13.01) | 1.06 (8.26)
  24-hour Diastolic Blood Pressure: number analyzed (Participants) | 68 | 66
  24-hour Diastolic Blood Pressure | 0.59 (6.08) | -0.73 (4.81)
  24-hour Mean Arterial Pressure: number analyzed (Participants) | 68 | 66
  24-hour Mean Arterial Pressure | 1.00 (8.20) | -0.14 (5.76)
  Sleep Systolic Blood Pressure: number analyzed (Participants) | 69 | 66
  Sleep Systolic Blood Pressure | 3.36 (16.65) | -0.21 (10.79)
  Sleep Diastolic Blood Pressure: number analyzed (Participants) | 69 | 66
  Sleep Diastolic Blood Pressure | 1.25 (8.81) | -0.51 (5.95)
  Sleep Mean Arterial Pressure: number analyzed (Participants) | 69 | 66
  Sleep Mean Arterial Pressure | 1.84 (10.79) | -0.37 (7.24)
  Wake Systolic Blood Pressure | 1.86 (12.08) | 1.42 (9.86)
  Wake Diastolic Blood Pressure | 0.51 (6.10) | -0.95 (5.79)
  Wake Mean Arterial Pressure | 0.81 (7.69) | -0.13 (6.42)
Statistical Analysis 1: Comparison: Control Arms (Pooled) vs Active Treatment Arms (Pooled); We conducted a linear mixed effects regression (LMER) to estimate the treatment effect of CPAP on mean 24hour Systolic Blood Pressure (SBP). Timepoint, treatment, and the timepoint* treatment interaction were included as fixed effects, as were randomization stratification factors. Subject was included as a random effect. Let: y = observed SBP; β = fixed effects; u = random effects; X = known design matrix; Z = vector of subjects Then our model is: y = Xβ + Zu + ε; Test type: Superiority or Other; Mean Difference (Net) = -2.677, 95% CI 2-sided [-5.915 to 0.561], Standard Error of Mean 1.652 — Presented average of the treatment effects on 24hr SBP at 6months and 12months: (6mo + 12mo)/ 2; Comparison: ActivePAP Control. Adjusted for randomization factors (CVD; site; sleepstudy type) with subjectspecific slopes and intercepts

2. Primary Outcome: Difference in CPAP Adherence by Active Treatment Arm
Description: Adherence to CPAP therapy was tracked remotely by modem transmission. Outcome reported is mean hours of PAP use per night at the 6-month timepoint. Comparison is between those with and without assignment to Motivational Enhancement as part of treatment randomization.
Time Frame: 6-months
Population: Intent to treat population for those assigned to Active PAP (all individuals who were randomized to one of the two PAP arms).
Measure: Mean (Standard Deviation); unit: hours/night
Groups:
- Active PAP With RT Support Only: Participants randomly assigned to either the Active PAP with RT Support arm (ActiveBeh).
- Active PAP With Motivational Enhancement: Participants randomly assigned to Active PAP with Behavioral Modification arm (Active+Beh).
Arm/Group | Active PAP With RT Support Only | Active PAP With Motivational Enhancement
Number analyzed (Participants) | 42 | 41
hours/night | 3.3 (2.7) | 4.4 (2.9)
Statistical Analysis 1: Comparison: Active PAP With RT Support Only vs Active PAP With Motivational Enhancement; We performed a mixed effects analysis of the effect of Motivational Enhancement (ME) on nightly CPAP adherence. Our model included every night of data and adjusted for intervention and study duration (number of nights), as well as randomization stratification factors (CVD; site; diagnostic sleepstudy type; PAP device type); Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Adjusted for intervention and study duration (number of nights), and randomization (CVD; site; diagnostic sleep study type; PAP device type); Mean Difference (Final Values) = 99 — Estimated value is minutes of use per night

3. Primary Outcome: Change From Baseline in 24-hour Blood Pressure at Months 6 and 12 (4 Arms)
Description: Blood pressure data was collected using a 24-hour ambulatory blood pressure monitor. Average of changes from baseline to 6 months and from baseline to 12 months.
Time Frame: Mean of 6- and 12-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) who had valid measurements of ambulatory blood pressure for baseline and at least one follow-up timepoint. Number analyzed differs between rows due to individuals having insufficient readings during wake and/or sleep.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 32 | 35 | 34
mmHg
  24-hour Systolic Blood Pressure: number analyzed (Participants) | 37 | 31 | 34 | 32
  24-hour Systolic Blood Pressure | 1.69 (13.17) | 1.96 (13.02) | 1.30 (8.75) | 0.80 (7.83)
  24-hour Diastolic Blood Pressure: number analyzed (Participants) | 37 | 31 | 34 | 32
  24-hour Diastolic Blood Pressure | 0.43 (6.78) | 0.77 (5.22) | -0.82 (4.82) | -0.63 (4.88)
  24-hour Mean Arterial Pressure: number analyzed (Participants) | 37 | 31 | 34 | 32
  24-hour Mean Arterial Pressure | 0.85 (8.81) | 1.17 (7.55) | -0.11 (5.98) | -0.16 (5.61)
  Sleep Systolic Blood Pressure: number analyzed (Participants) | 37 | 32 | 34 | 32
  Sleep Systolic Blood Pressure | 2.1 (17.84) | 4.81 (15.32) | -1.02 (12.08) | 0.65 (9.36)
  Sleep Diastolic Blood Pressure: number analyzed (Participants) | 37 | 32 | 34 | 32
  Sleep Diastolic Blood Pressure | 0.51 (9.08) | 2.1 (8.55) | -0.88 (6.58) | -0.12 (5.27)
  Sleep Mean Arterial Pressure: number analyzed (Participants) | 37 | 32 | 34 | 32
  Sleep Mean Arterial Pressure | 0.93 (11.87) | 2.89 (9.46) | -0.74 (8.23) | 0.02 (6.13)
  Wake Systolic Blood Pressure | 1.83 (13.65) | 1.89 (10.18) | 1.69 (10.64) | 1.14 (9.14)
  Wake Diastolic Blood Pressure | 0.75 (7.08) | 0.24 (4.84) | -1.06 (6.22) | -0.83 (5.42)
  Wake Mean Arterial Pressure | 0.73 (9.04) | 0.91 (5.90) | -0.15 (7.20) | -0.10 (5.63)

4. Primary Outcome: Change From Baseline in 24-hour Blood Pressure at Month 12 by Pooled Arms
Description: Blood pressure data was collected using a 24-hour ambulatory blood pressure monitor. The 2 Active arms and 2 Control arms were pooled to create a 2-arm analysis. Outcome reported is change from baseline to 12-months. Control arms and Active arms were pooled, respectively, for analysis.
Time Frame: 12-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) who had valid measurements of ambulatory blood pressure for baseline and 12 Month follow-up. Number analyzed differs between rows due to individuals having insufficient readings during wake and/or sleep.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Arms (Pooled) | Active Treatment Arms (Pooled)
Number analyzed (Participants) | 40 | 35
mmHg
  24-hour Systolic Blood Pressure: number analyzed (Participants) | 38 | 33
  24-hour Systolic Blood Pressure | 0.37 (16.52) | 0.17 (8.95)
  24-hour Diastolic Blood Pressure: number analyzed (Participants) | 38 | 33
  24-hour Diastolic Blood Pressure | -0.22 (6.48) | -1.57 (5.12)
  24-hour Mean Arterial Pressure: number analyzed (Participants) | 38 | 33
  24-hour Mean Arterial Pressure | -0.03 (9.33) | -0.99 (6.15)
  Sleep Systolic Blood Pressure: number analyzed (Participants) | 39 | 34
  Sleep Systolic Blood Pressure | 2.61 (21.74) | -1.09 (14.31)
  Sleep Diastolic Blood Pressure: number analyzed (Participants) | 39 | 34
  Sleep Diastolic Blood Pressure | 0.57 (10.02) | -1.39 (7.87)
  Sleep Mean Arterial Pressure: number analyzed (Participants) | 39 | 34
  Sleep Mean Arterial Pressure | 0.83 (12.79) | -1.10 (9.57)
  Wake Systolic Blood Pressure | -0.71 (16.60) | -0.40 (11.82)
  Wake Diastolic Blood Pressure | -0.78 (6.90) | -2.16 (6.82)
  Wake Mean Arterial Pressure | -0.80 (9.75) | -1.16 (7.61)

5. Primary Outcome: Change From Baseline in 24-hour Blood Pressure at Month 6 by Pooled Arms
Description: Blood pressure data was collected using a 24-hour ambulatory blood pressure monitor. The 2 Active arms and 2 Control arms were pooled to create a 2-arm analysis. Outcome reported mean change from baseline to 6-months. Control arms and Active arms were pooled, respectively, for analysis.
Time Frame: 6-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) who had valid measurements of ambulatory blood pressure for baseline and 6 Month follow-up. Number analyzed differs between rows due to individuals having insufficient readings during wake and/or sleep.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Arms (Pooled) | Active Treatment Arms (Pooled)
Number analyzed (Participants) | 64 | 66
mmHg
  24-hour Systolic Blood Pressure: number analyzed (Participants) | 59 | 64
  24-hour Systolic Blood Pressure | 2.60 (9.90) | 1.24 (8.78)
  24-hour Diastolic Blood Pressure: number analyzed (Participants) | 59 | 64
  24-hour Diastolic Blood Pressure | 0.97 (5.50) | -0.53 (5.16)
  24-hour Mean Arterial Pressure: number analyzed (Participants) | 59 | 64
  24-hour Mean Arterial Pressure | 1.52 (6.80) | 0.06 (6.14)
  Sleep Systolic Blood Pressure: number analyzed (Participants) | 61 | 64
  Sleep Systolic Blood Pressure | 4.58 (14.28) | -0.18 (10.64)
  Sleep Diastolic Blood Pressure: number analyzed (Participants) | 61 | 64
  Sleep Diastolic Blood Pressure | 2.07 (8.20) | -0.27 (6.01)
  Sleep Mean Arterial Pressure: number analyzed (Participants) | 61 | 64
  Sleep Mean Arterial Pressure | 2.94 (9.41) | -0.30 (7.19)
  Wake Systolic Blood Pressure: number analyzed (Participants) | 63 | 66
  Wake Systolic Blood Pressure | 2.84 (11.05) | 2.10 (10.31)
  Wake Diastolic Blood Pressure: number analyzed (Participants) | 63 | 66
  Wake Diastolic Blood Pressure | 0.93 (6.25) | -0.61 (6.04)
  Wake Mean Arterial Pressure: number analyzed (Participants) | 63 | 66
  Wake Mean Arterial Pressure | 1.42 (7.31) | 0.29 (6.78)

6. Primary Outcome: Change From Baseline in 24-hour Blood Pressure at Month 12 (4 Arms)
Description: Blood pressure data was collected using a 24-hour ambulatory blood pressure monitor. Outcome reported is mean change from baseline to 12-months.
Time Frame: 12-months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 22 | 18 | 18 | 17
mmHg
  24-hour Systolic Blood Pressure: number analyzed (Participants) | 22 | 16 | 17 | 16
  24-hour Systolic Blood Pressure | -0.97 (15.36) | 2.22 (18.36) | -0.09 (10.42) | 0.45 (7.41)
  24-hour Diastolic Blood Pressure: number analyzed (Participants) | 22 | 16 | 17 | 16
  24-hour Diastolic Blood Pressure | -0.68 (7.32) | 0.40 (5.29) | -1.61 (5.00) | -1.53 (5.40)
  24-hour Mean Arterial Pressure: number analyzed (Participants) | 22 | 16 | 17 | 16
  24-hour Mean Arterial Pressure | -0.78 (9.90) | 1.01 (8.68) | -1.10 (6.64) | -0.87 (5.78)
  Sleep Systolic Blood Pressure: number analyzed (Participants) | 22 | 17 | 18 | 16
  Sleep Systolic Blood Pressure | 0.40 (22.7) | 5.48 (20.82) | -3.79 (17.02) | 1.94 (10.17)
  Sleep Diastolic Blood Pressure: number analyzed (Participants) | 22 | 17 | 18 | 16
  Sleep Diastolic Blood Pressure | -0.52 (10.47) | 1.97 (9.53) | -2.54 (9.17) | -0.11 (6.12)
  Sleep Mean Arterial Pressure: number analyzed (Participants) | 22 | 17 | 18 | 16
  Sleep Mean Arterial Pressure | -0.51 (14.00) | 2.57 (11.21) | -2.88 (11.44) | 0.91 (6.71)
  Wake Systolic Blood Pressure | -1.91 (14.84) | 0.74 (18.87) | -0.75 (15.15) | -0.02 (7.27)
  Wake Diastolic Blood Pressure | -0.91 (7.60) | -0.62 (6.15) | -2.25 (8.00) | -2.06 (5.55)
  Wake Mean Arterial Pressure | -1.44 (10.54) | -0.005 (8.92) | -1.59 (9.91) | -0.71 (4.28)

7. Primary Outcome: Change From Baseline in 24-hour Blood Pressure at Month 6 (4 Arms)
Description: Blood pressure data was collected using a 24-hour ambulatory blood pressure monitor. Outcome reported is mean change from baseline to 6-months.
Time Frame: 6-months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 34 | 30 | 34 | 32
mmHg
  24-hour Systolic Blood Pressure: number analyzed (Participants) | 31 | 28 | 33 | 31
  24-hour Systolic Blood Pressure | 2.45 (10.77) | 2.77 (9.04) | 2.12 (8.94) | 0.29 (8.65)
  24-hour Diastolic Blood Pressure: number analyzed (Participants) | 31 | 28 | 33 | 31
  24-hour Diastolic Blood Pressure | 0.85 (6.08) | 1.11 (4.89) | -0.40 (5.15) | -0.67 (5.24)
  24-hour Mean Arterial Pressure: number analyzed (Participants) | 31 | 28 | 33 | 31
  24-hour Mean Arterial Pressure | 1.38 (7.53) | 1.67 (6.01) | 0.44 (6.23) | -0.35 (6.12)
  Sleep Systolic Blood Pressure: number analyzed (Participants) | 32 | 29 | 33 | 31
  Sleep Systolic Blood Pressure | 3.67 (12.37) | 5.59 (16.29) | -0.21 (11.91) | -0.15 (9.30)
  Sleep Diastolic Blood Pressure: number analyzed (Participants) | 32 | 29 | 33 | 31
  Sleep Diastolic Blood Pressure | 1.53 (7.09) | 2.65 (9.37) | -0.21 (6.51) | -0.34 (5.53)
  Sleep Mean Arterial Pressure: number analyzed (Participants) | 32 | 29 | 33 | 31
  Sleep Mean Arterial Pressure | 2.34 (8.75) | 3.60 (10.20) | -0.10 (8.08) | -0.50 (6.22)
  Wake Systolic Blood Pressure: number analyzed (Participants) | 33 | 30 | 34 | 32
  Wake Systolic Blood Pressure | 3.31 (13.20) | 2.33 (8.26) | 3.14 (10.02) | 0.99 (10.67)
  Wake Diastolic Blood Pressure: number analyzed (Participants) | 33 | 30 | 34 | 32
  Wake Diastolic Blood Pressure | 1.46 (7.26) | 0.36 (4.96) | -0.50 (6.14) | -0.72 (6.02)
  Wake Mean Arterial Pressure: number analyzed (Participants) | 33 | 30 | 34 | 32
  Wake Mean Arterial Pressure | 1.77 (8.81) | 1.04 (5.34) | 0.70 (6.97) | -0.13 (6.65)

8. Secondary Outcome: Change in 36-Item Short Form Survey (SF-36) Measures (4 Arm)
Description: The 36-Item Short Form Survey (SF-36) is a patient-reported survey of patient health. The SF-36 scores range from 0-100, with lower scores indicating greater disability. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) with valid measurements of ambulatory blood pressure for baseline and at least one follow-up timepoint. Not all measures were able to be collected from all participants. Not all participants completed 12 month visits (due to randomization date).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 32 | 36 | 34
units on a scale
  SF-36 Physical Component: number analyzed (Participants) | 38 | 32 | 35 | 32
  SF-36 Physical Component | -1.3 (7.3) | -1.3 (6.4) | 1.1 (4.7) | 1.8 (4.7)
  SF-36 Mental Component: number analyzed (Participants) | 38 | 32 | 35 | 32
  SF-36 Mental Component | 0.6 (7.6) | 2.9 (6.4) | 3.9 (8.4) | 2.2 (6.3)
  SF-36 Vitality Subscale: number analyzed (Participants) | 38 | 32 | 36 | 33
  SF-36 Vitality Subscale | 0.9 (14.3) | 5.6 (11.4) | 12.7 (14.9) | 6.4 (12.6)
  SF-36 Physical Functioning | -1.8 (16.5) | 0.4 (14.4) | 3.3 (11.2) | 3.1 (13.9)
  SF-36 Bodily Pain | -1.7 (18.8) | -3.4 (23.2) | 4.1 (14.4) | 7.8 (19.4)
  SF-36 General Health Perceptions: number analyzed (Participants) | 38 | 32 | 35 | 34
  SF-36 General Health Perceptions | -4.4 (17.2) | -0.04 (15.8) | 5.0 (12.6) | 7.1 (14.6)
  SF-36 Physical Role Functioning | -2.2 (21.3) | -0.9 (22.2) | 3.4 (15.9) | -2.11 (17.3)
  SF-36 Emotional Role Functioning: number analyzed (Participants) | 38 | 32 | 36 | 33
  SF-36 Emotional Role Functioning | 0 (20.1) | 9.2 (27.1) | 3.7 (19.5) | 5.2 (22.4)
  SF-36 Social Role Functioning | 1.8 (17.7) | 0.4 (14.1) | 4.5 (15.4) | 3.7 (14.1)
  SF-36 Mental Health: number analyzed (Participants) | 38 | 32 | 36 | 33
  SF-36 Mental Health | -0.5 (13.4) | 1.1 (9.1) | 6.1 (15.6) | 1.1 (11.5)

9. Secondary Outcome: Change in Epworth Sleepiness Scale (ESS) (4 Arm)
Description: The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness. The ESS score ranges from 0 - 24, with higher scores indicating increasing possibility of specific sleep disorders. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 32 | 36 | 34
units on a scale | -0.6 (3.1) | -1.0 (3.3) | -1.9 (3.1) | -1.6 (4.0)

10. Secondary Outcome: Change in Patient Health Questionnaire (PHQ8) (4 Arm)
Description: The Patient Health Questionnaire (PHQ-8) is a scale intended to measure depression. The PHQ-8 score ranges from 0 24, with higher scores indicating increasing severity of depression. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 32 | 35 | 33
units on a scale | -0.4 (3.2) | -0.9 (2.5) | -1.7 (3.9) | -1.4 (4.0)

11. Secondary Outcome: Change in the Calgary Sleep Apnea Quality of Life Index (SAQLI) (4 Arm)
Description: The Calgary Sleep Apnea Quality of Life Index (SAQLI) is a scale intended to measure disease-specific quality of life. The SAQLI score ranges from 1 - 7, with higher scores indicating a higher quality of life. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 32 | 36 | 33
units on a scale | 0.1 (0.4) | 0.2 (0.6) | -0.1 (0.7) | -0.1 (0.7)

12. Secondary Outcome: Change in C-Reactive Protein at Months 6 and 12 (4 Arm)
Description: C-Reactive Protein laboratory measurements were calculated from blood samples collected through fasting phlebotomy. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 34 | 35 | 33
mg/L
  InCRP | 0.2 (0.6) | -0.02 (0.8) | 0.0003 (0.6) | 0.2 (0.5)
  InCRP (excluding raw >10): number analyzed (Participants) | 35 | 32 | 31 | 31
  InCRP (excluding raw >10) | 0.2 (0.6) | 0.1 (0.6) | 0.1 (0.5) | 0.1 (0.5)

13. Secondary Outcome: Change in Lipid Panel at 6 and 12 Months (4 Arm)
Description: Lipid panel measurements were calculated from blood samples collected through fasting phlebotomy. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) with valid measurements of ambulatory blood pressure for baseline and at least one follow-up timepoint. Lipid measures were not able to be collected from all participants. Not all participants completed 12 month visits (due to randomization date).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 34 | 35 | 33
mg/dL
  Triglycerides | 9.4 (56.9) | 1.5 (47.1) | 4.0 (37.3) | 1.8 (28.8)
  HDL Cholesterol | -0.5 (5.2) | 1.7 (6.8) | -0.7 (7.8) | -0.05 (5.2)
  LDL Cholesterol: number analyzed (Participants) | 37 | 34 | 35 | 33
  LDL Cholesterol | 5.1 (17.5) | 2.5 (20.5) | 1.4 (16.5) | 6.0 (19.0)
  Total Cholesterol | 5.6 (19.5) | 4.5 (27.3) | 0.7 (19.5) | 6.3 (20.6)
  VLDL Cholesterol: number analyzed (Participants) | 37 | 34 | 35 | 33
  VLDL Cholesterol | 0.3 (5.7) | 0.2 (9.5) | 0.1 (8.0) | 0.2 (5.8)

14. Secondary Outcome: Change in Glucose, Fibrinogen, Creatinine and BNP at Months 6 and 12 (4 Arm)
Description: Glucose, Fibrinogen, Creatinine and BNP measurements were calculated from blood and urine samples collected through fasting phlebotomy and urine collection. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 34 | 35 | 33
mg/dL
  Glucose | 2.9 (16.2) | 3.9 (47.1) | 10.9 (45.9) | 1.0 (12.3)
  Fibrinogen: number analyzed (Participants) | 35 | 34 | 30 | 30
  Fibrinogen | 18.9 (56.3) | -2.0 (72.7) | 2.75 (45.5) | 11.9 (63.8)
  Urine Creatinine: number analyzed (Participants) | 38 | 34 | 33 | 31
  Urine Creatinine | -7.8 (62.9) | -9.5 (66.1) | 8.7 (50.5) | -5.4 (41.0)
  Serum Creatinine: number analyzed (Participants) | 34 | 33 | 32 | 31
  Serum Creatinine | -0.007 (0.1) | -0.01 (0.1) | -0.01 (0.1) | 0.007 (0.1)
  B-type Natriuretic Peptide (BNP): number analyzed (Participants) | 34 | 33 | 31 | 31
  B-type Natriuretic Peptide (BNP) | -34.3 (111.6) | 4.7 (138.7) | 19.1 (175.1) | -3.3 (68.7)

15. Secondary Outcome: Change From Baseline in Hemoglobin A1c Percentage at Months 6 and 12 (4 Arm)
Description: Hemoglobin A1c percentage was calculated from blood samples collected through fasting phlebotomy. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage glycosylated hemoglobin
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 33 | 34 | 32
percentage glycosylated hemoglobin | 0.1 (0.4) | -0.2 (0.6) | -0.04 (0.5) | 0.1 (0.4)

16. Secondary Outcome: Change From Baseline in Fasting Insulin at Months 6 and 12 (4 Arm)
Description: Fasting Insulin was calculated from blood samples collected through fasting phlebotomy. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 33 | 36 | 32
uIU/mL | -0.9 (6.7) | 2.8 (12.0) | -2.4 (15.4) | 1.1 (5.9)

17. Secondary Outcome: Change in Interleukin 6 (IL-6) at Months 6 and 12 (4 Arm)
Description: Interleukin 6 (IL-6) was calculated from blood samples collected through fasting phlebotomy. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pg/dL
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 32 | 36 | 32
pg/dL | 5.3 (30.2) | 0.5 (2.7) | -2.5 (15.6) | 0.4 (2.1)

18. Secondary Outcome: Change in Glomerular Filtration Rate (GFR) at Months 6 and 12 (4 Arm)
Description: Glomerular Filtration Rate was calculated from blood samples collected through fasting phlebotomy. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 34 | 33 | 32 | 31
mL/min/1.73m^2 | -0.2 (9.9) | 0.6 (11.0) | 0.007 (8.3) | -1.15 (9.1)

19. Secondary Outcome: Change in Urine Microalbumin at Months 6 and 12 (4 Arm)
Description: Urine Microalbumin was calculated from urine samples. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 34 | 33 | 31
ug/mL | -16.7 (31.2) | 45.4 (315.7) | 3.7 (43.0) | 8.2 (58.2)

20. Secondary Outcome: Change in Urinary Albumin Creatinine Ratio at Months 6 and 12 (4 Arm)
Description: Urinary Albumin Creatinine Ratio was calculated from urine samples. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ug/mg
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 34 | 33 | 31
ug/mg | -9.3 (29.4) | 84.6 (568.0) | 1.2 (55.9) | 6.0 (58.8)

21. Secondary Outcome: Change in Plasminogen Activator Inhibitor-1 (PAI-1) at Months 6 and 12 (4 Arm)
Description: Plasminogen Activator Inhibitor-1 (PAI-1) was calculated from blood samples. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: AU/mL
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 33 | 35 | 32
AU/mL | 0.8 (2.5) | 0.2 (3.7) | 1.1 (6.9) | 0.3 (4.0)

22. Secondary Outcome: Change in Pulse Wave Velocity (PWV) at Months 6 and 12 (4 Arms)
Description: Tonometry measurements of arterial stiffness were collected using a Sphygmacor. Outcome reported is mean of change from baseline to 6-months and baseline to 12-months.
Time Frame: Mean of 6- and 12-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) with valid measurements of ambulatory blood pressure for baseline and at least one follow-up timepoint. Tonometry measures were not able to be collected from all participants. Not all participants completed 12 month visits (due to randomization date).
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 27 | 26 | 31 | 24
m/s | 0.05 (1.9) | -0.03 (1.5) | -0.2 (2.0) | 0.1 (1.1)

23. Secondary Outcome: Change in Augmentation Index at Months 6 and 12 (4 Arms)
Description: as for outcome 22
Time Frame: Mean of 6- and 12-months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent of central pulse pressure
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 35 | 28 | 31 | 29
percent of central pulse pressure | -1.2 (9.2) | -0.4 (8.0) | 0.9 (7.5) | -0.9 (8.0)

24. Secondary Outcome: Left Ventricular (LV) Mass Index (4 Arm) - Baseline
Description: Baseline Left Ventricular Mass Index measured via echocardiography.
Time Frame: 12-months
Population: Intent to treat population (all individuals who were randomized to a treatment arm) with valid measurements of ambulatory blood pressure for baseline and at least one follow-up timepoint. Echocardiography measures were not able to be collected from all participants. Not all participants completed 12 month visits (due to randomization date).
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 37 | 37 | 39 | 37
g/m2 | 82.4 (15.7) | 78.5 (16.4) | 77.0 (19.0) | 76.3 (18.9)

25. Secondary Outcome: Left Atrial (LA) Volume Index (4 Arm) - Baseline
Description: Baseline Left Atrial Mass Index measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: m/m2
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 37 | 39 | 37
m/m2 | 27.1 (11.0) | 25.3 (10.6) | 25.1 (6.9) | 24.2 (7.7)

26. Secondary Outcome: End-Diastolic Volume (4 Arm) - Baseline
Description: Baseline End-Diastolic Volume measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 37 | 38 | 37
cm | 113.8 (18.2) | 111.8 (19.8) | 113.4 (22.8) | 112.3 (19.7)

27. Secondary Outcome: Ejection Fraction (4 Arm) - Baseline
Description: Baseline Ejection Fraction measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 37 | 38 | 37
percent ejection fraction | 60.2 (4.1) | 60.9 (2.7) | 60.8 (6.6) | 59.9 (4.6)

28. Secondary Outcome: Right Ventricular Fractional Area Change (4 Arm) - Baseline
Description: Baseline RV Fractional Area Change measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percentage change in RV area
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 35 | 34 | 33 | 36
percentage change in RV area | 0.5 (0.1) | 0.5 (0.0) | 0.5 (0.1) | 0.5 (0.0)

29. Secondary Outcome: Tricuspid Annular Peak Systolic Myocardial Velocity (4 Arm) - Baseline
Description: Baseline Tricuspid Annular Peak Systolic Myocardial Velocity measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 34 | 35 | 38 | 34
cm/sec | 14.2 (3.5) | 13.1 (3.0) | 13.5 (2.4) | 13.1 (3.1)

30. Secondary Outcome: Pulmonary Vascular Resistance (4 Arm) - Baseline
Description: Baseline Pulmonary Vascular Resistance measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Wood units
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 22 | 19 | 22 | 20
Wood units | 154.6 (30.1) | 135.5 (40.3) | 151.1 (35.2) | 157.0 (39.1)

31. Secondary Outcome: E/Em Lateral Ratio (4 Arm) - Baseline
Description: Baseline E/Em Lateral Ratio measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mitral velocity ratio (absolute units)
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 38 | 36 | 39 | 36
mitral velocity ratio (absolute units) | 8.6 (3.4) | 8.3 (2.7) | 8.4 (2.7) | 7.9 (2.5)

32. Secondary Outcome: Peak Tricuspid Regurgitation Velocity (4 Arm) - Baseline
Description: Baseline Peak Tricuspid Regurgitation Velocity measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 23 | 21 | 23 | 21
cm/sec | 243.5 (22.1) | 240.4 (23.9) | 244.0 (21.3) | 248.3 (30.7)

33. Secondary Outcome: Left Ventricular Mass Index (4 Arm) - 12 Month
Description: Endpoint Left Ventricular Mass Index measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 22 | 17 | 15 | 16
g/m2 | 82.1 (17.3) | 76.9 (15.6) | 74.2 (23.7) | 70.4 (18.0)

34. Secondary Outcome: Left Atrial Volume Index (4 Arm) - 12 Month
Description: Endpoint Left Atrial Volume Index measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: m/m2
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 22 | 17 | 15 | 16
m/m2 | 25.5 (11.7) | 22.3 (6.7) | 24.6 (6.4) | 20.7 (5.6)

35. Secondary Outcome: End-Diastolic Volume (4 Arm) - 12 Month
Description: Endpoint End-Diastolic Volume measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 22 | 17 | 16 | 16
cm | 110.7 (17.4) | 112.3 (19.6) | 115.5 (26.9) | 106.1 (14.0)

36. Secondary Outcome: Ejection Fraction (4 Arm) - 12 Month
Description: Endpoint Ejection Fraction measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percentage ejection fraction
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 22 | 17 | 16 | 16
percentage ejection fraction | 61.1 (4.7) | 61.4 (4.2) | 60.6 (5.1) | 60.9 (2.7)

37. Secondary Outcome: Right Ventricular Fractional Area Change (4 Arm) - 12 Month
Description: Endpoint Right Ventricular Fractional Area Change measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: percentage change in RV area
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 21 | 14 | 16 | 15
percentage change in RV area | 0.5 (0.0) | 0.5 (0.0) | 0.5 (0.0) | 0.5 (0.0)

38. Secondary Outcome: Tricuspid Annular Peak Systolic Myocardial Velocity (4 Arm) - 12 Month
Description: Endpoint Tricuspid Annular Peak Systolic Myocardial Velocity measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 21 | 17 | 16 | 15
cm/sec | 14.1 (3.6) | 13.5 (2.5) | 13.6 (2.5) | 14.1 (2.5)

39. Secondary Outcome: Pulmonary Vascular Resistance (4 Arm) - 12 Month
Description: Endpoint Pulmonary Vascular Resistance measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Wood units
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 14 | 7 | 8 | 9
Wood units | 148.4 (26.7) | 138.2 (16.6) | 144.0 (54.8) | 131.3 (29.1)

40. Secondary Outcome: E/Em Lateral Ratio (4 Arm) - 12 Month
Description: Endpoint E/Em Lateral Ratio measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mitral velocity ratio (absolute units)
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 22 | 17 | 16 | 16
mitral velocity ratio (absolute units) | 8.8 (3.2) | 8.2 (2.5) | 9.2 (2.9) | 8.4 (2.8)

41. Secondary Outcome: Peak Tricuspid Regurgitation Velocity (4 Arm) - 12 Month
Description: 12 Month Peak Tricuspid Regurgitation Velocity measured via echocardiography.
Time Frame: 12-months
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Number analyzed (Participants) | 14 | 7 | 8 | 10
cm/sec | 235.4 (32.9) | 253.1 (35.0) | 232.0 (13.6) | 254.7 (23.3)

ADVERSE EVENTS:
Time Frame: 6 months to 1 year, depending on participant's randomization date.
Description: Adverse events were reported to study coordinator during bimonthly phone assessments. Adverse events that were reported to other staff members on treatment visits (respiratory and/or behavioral therapist) or study visits were reported to the study coordinator.
Groups:
- Sham PAP (Sham): In addition to receiving CMT and active-PAP, participants will meet with a behavioral interventionist in addition to PAP-specialist visits. Participants also would speak with the behavioral interventionist over the course of the study (set up, 1-week, 3-week, 1-month, 2-months, 3-months, 5-months and 8-months). The duration of the first 2 behavioral intervention sessions are estimated to be 1-hour long, with subsequent 30-minutes intervention sessions. The intervention will be based on social cognitive theory and feedback concerning adherence with targeted problem solving training.
- Active PAP With RT Support (Active-Beh): In addition to receiving CMT, participants in this treatment arm will receive a sham PAP unit. Sham devices look like active PAP devices, however, the exhalation port is increased and an orifice-resistor is inserted between the pump and tubing, creating a marginal pressure. A heated humidifier will be provided with this device and PAP masks will be fit and provided following the same procedures as for the active-PAP arms.
- Active PAP With Behavioral Modification (Active+Beh): In addition to receiving CMT, participants will receive active-PAP and meet with a PAP-specialist . The PAP specialist would meet with the participant in person throughout the course of the study (set-up, 1-week, 1-month, 3-month, 6-month, and 9-month). Using the available data from the PAP monitor, the PAP specialist will discuss PAP use, mask leaks, and residual AHI to assist with troubleshooting. Adjustments to equipment would be performed as needed to improve adherence. It is estimated that each in-person follow-up adherence visit with the PAP-specialist would last 30 minutes.
Arm/Group | Conservative Medical Therapy (CMT) | Sham PAP (Sham) | Active PAP With RT Support (Active-Beh) | Active PAP With Behavioral Modification (Active+Beh)
Serious Adverse Events (participants affected / at risk) | 7/44 | 5/42 | 2/42 | 4/41
Other Adverse Events (participants affected / at risk) | 17/44 | 22/42 | 16/42 | 18/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conservative Medical Therapy (CMT) (N=44) | Sham PAP (Sham) (N=42) | Active PAP With RT Support (Active-Beh) (N=42) | Active PAP With Behavioral Modification (Active+Beh) (N=41)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar Ischemia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombotic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Breast Abscess (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysponea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Bacterial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic Dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conservative Medical Therapy (CMT) (N=44) | Sham PAP (Sham) (N=42) | Active PAP With RT Support (Active-Beh) (N=42) | Active PAP With Behavioral Modification (Active+Beh) (N=41)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dysponea (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 4 (5) | 4 (4) | 2 (2) | 3 (3)
Oedema Peripheral (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Dermatitis Allergic (Immune system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Urticaria (Immune system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blood pressure increased (Investigations) | 4 (4) | 5 (6) | 3 (3) | 4 (4)
Athralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Prostate Cancer (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 1 (2) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Carpal Tunnel Decompression (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No